CLINICAL TRIAL: NCT03684564
Title: Rivaroxaban Versus Warfarin for Stroke Patients With Antiphospholipid Syndrome, With or Without SLE (RISAPS): a Randomised, Controlled, Open-label, Phase IIb, Non-inferiority Proof of Principle Trial.
Brief Title: RIvaroxaban for Stroke Patients With AntiPhospholipid Syndrome
Acronym: RISAPS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other); Barking, Havering and Redbridge University Hospitals NHS Trust (Other); Hammersmith Hospitals NHS Trust (Other); Epsom and St Helier University Hospitals NHS Trust (Other); Barts & The London NHS Trust (Other); King's College Hospital NHS Trust (Other); Versus Arthritis (Funder) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTU/2015/174
Record Dates: First submitted 2018-08-13; First posted 2018-09-25 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Antiphospholipid Syndrome; Systemic Lupus Erythematosus; Stroke; Ischemic Stroke; Brain Ischemia
MeSH Terms: conditions — Antiphospholipid Syndrome; Lupus Erythematosus, Systemic; Stroke; Ischemic Stroke; Brain Ischemia | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Intervention Model Description: Participants enrolled in RISAPS will be randomly allocated 1:1 to receive either oral rivaroxaban 15mg twice daily or oral warfarin (standard of care in the RISAPS trial) to maintain a target INR of 3.5 (range 3.0-4.0) for 24 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Treatment Arm) (Experimental)
  Interventions: Drug: Rivaroxaban
- Warfarin (Control Arm) (Active Comparator)
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban — Oral tablet 15 mg twice daily for 24 months
  Arms: Rivaroxaban (Treatment Arm)
Drug: Warfarin — Oral anticoagulant given as standard of care in the RISAPS trial to maintain a target INR of 3.5 (range 3.0-4.0) for 24 months
  Arms: Warfarin (Control Arm)

SUMMARY:
Rivaroxaban versus warfarin for stroke patients with antiphospholipid syndrome, with or without SLE (RISAPS): a randomised, controlled, open-label, phase IIb, non-inferiority proof of principle trial.

40 patients will be randomised with a ratio of 1:1 to receive either:

* Rivaroxaban 15mg twice daily orally for 24 months or
* Warfarin (standard of care in the RISAPS trial) to maintain a target INR of 3.5 (range 3.0-4.0) for 24 months.

The primary outcome of the trial is the rate of change in brain white matter hyperintensity (WMH) volume between baseline and 24 months follow up, assessed on brain magnetic resonance imaging (MRI), a surrogate marker of ischaemic damage.

DETAILED DESCRIPTION:
The RISAPS trial follows on from the RAPS (Rivaroxaban in Antiphospholipid Syndrome) study that showed that rivaroxaban could offer a potentially effective alternative to warfarin for patients with antiphospholipid syndrome (APS) who have thrombosis (blood clots) in their veins, rather than in their arteries and require standard intensity anticoagulation (blood thinning).

Currently, APS patients who have had an ischaemic stroke (which occurs when blood flow to an area of brain is cut off) are treated with warfarin to reduce the risk of a recurrence. Warfarin tends to have a variable 'blood thinning' effect in patients with APS, necessitating frequent (usually weekly) INR blood tests to monitor the effect of the warfarin, which is inconvenient for patients.

The RISAPS trial will compare higher intensity (higher dose) rivaroxaban versus higher intensity warfarin (current standard of care treatment) for 24 months, in APS patients, with or without lupus (systemic lupus erythematosus; SLE), requiring higher intensity anticoagulation after experiencing a stroke, a 'mini stroke' (also known as a transient ischaemic attack) or other ischaemic brain damage (caused by blood clots in the brain arteries or smaller blood vessels). When compared with warfarin, a dvantages of rivaroxaban include, fixed dose prescribing and no need for monitoring of anticoagulant effect.

Furthermore, rivaroxaban has fewer drug-food interactions, and significantly fewer drug-drug interactions than warfarin. If rivaroxaban is no worse than warfarin for anticoagulation of APS patients with stroke or other ischaemic brain manifestations, it could become the standard of care for the treatment of APS patients, with or without lupus, who have experienced stroke or other ischaemic brain manifestations and improve patients' quality of life.

ELIGIBILITY:
Inclusion Criteria

1. Patients must be confirmed as having persistent antiphospholipid antibodies (aPL), defined as: positivity of one or more aPL, i.e. lupus anticoagulant, IgG and/or IgM anticardiolipin and/or anti beta 2 glycoprotein I antibodies at >40 GPL or MPL units or > the 99th centile of normal, on two or more occasions, at least 12 weeks apart. See Appendix 3 and Exclusion criteria for more information.
2. One or more of: a) Ischaemic stroke; b) transient ischaemic attack (TIA) with evidence of either acute or chronic ischaemic injury on brain magnetic resonance imaging (MRI) (including diffusion-weighted magnetic resonance imaging (DWI) lesion(s), previous cortical or subcortical infarction(s), or white matter hyperintensities) and diagnosed by a clinician with expertise in stroke; c) brain infarcts (territorial or subcortical) or white matter hyperintensities (WMH) of presumed vascular origin on brain MRI, with or without cognitive impairment; and an expert clinical opinion that anticoagulation is a reasonable treatment option (with the aim of preventing ischaemic brain injury).
3. Patients must weigh ≥ 50kg and ≤ 135kg.
4. Women must be on adequate contraception, barrier or hormonal, unless postmenopausal or sterilised.

Exclusion Criteria

1. Patients who are triple positive for antiphospholipid antibodies (presence of lupus anticoagulant, IgG and/or IgM anticardiolipin and anti beta 2 glycoprotein I antibodies at >40 GPL or MPL units or > the 99th centile of normal*.

   (*patients who have previously been triple aPL-positive and have single or double aPL positivity on at least 2 occasions over at least 6 months, including once within 1 month prior to randomisation, can be recruited to the trial)
2. Pregnant or lactating women
3. Severe renal impairment with creatinine clearance < 30 mL/min (i.e. 29 mL/min or less)
4. Liver function tests ALT > 3 x ULN
5. Cirrhotic patients with Child Pugh B or C
6. Thrombocytopenia (platelets < 75 x 109/L)
7. Non-adherence on warfarin (based on clinical assessment)
8. Patients taking strong inhibitors of both CYP3A4 and P-gp pathways such as

   1. Systemic azole antifungals (e.g. ketoconazole, itraconazole, voriconazole, posaconazole)
   2. Patients on human immunodeficiency virus (HIV) protease inhibitors (e.g. ritonavir)
9. Patients on strong CYP3A4 inducers (e.g. rifampicin, phenytoin, carbamazepine, phenobarbital or St. John's Wort)
10. Patients on dronedarone
11. Patients on levetiracetam, sodium valproate/valproic acid, oxcarbazepine or topiramate
12. Patients less than 18 years of age
13. Refusal to consent to the site informing General Practitioner (GP) and Healthcare Professional responsible for anticoagulation care of the participant.
14. Contraindications to MRI (e.g. cardiac pacemaker, severe claustrophobia, inability to lie flat: patients who do not meet local safety rules for MRI).
15. Patients at high risk of bleeding and not suitable for anticoagulation therapy.
16. Previous known allergy or intolerance to warfarin or rivaroxaban.
17. Women planning to become pregnant within the 2-year follow-up period.
18. Patients with known galactose intolerance, total lactase deficiency or galactose malabsorption.
19. Patients who have had active cancer (excluding non-melanoma skin cancers) within the last 2 years
20. Any other reason that the PI or delegate considers would make the patient unsuitable to enter RISAPS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
To compare the efficacy of high-intensity oral rivaroxaban (15mg twice daily) vs high-intensity warfarin, target INR 3.5 (range 3.0-4.0), in patients with APS with or without SLE who have had a stroke or other ischaemic brain manifestations. | 24 months
  The comparison of efficacy will be based on the rate of change in brain white matter hyperintensity (WMH) volume on MRI, a surrogate marker of ischaemic damage, between baseline and 24 months follow up.

SECONDARY OUTCOMES:
A) Efficacy - Neuroradiological markers | 24 months
  i) Mean diffusivity and fractional anisotropy as a measure of microstructural white matter damage derived from diffusion tensor imaging (DTI) ii) Changes in total brain volume, white matter volume and grey matter volume on T1 weighted volumetric images iii) Brain infarcts
  1. cortical or subcortical
  2. assessment of volume iv) Cerebral venous occlusions
Clinical | 24 months
  (i) Vascular events
  1. Ischaemic stroke or transient ischaemic attack
  2. Occlusive arterial events in other sites including systemic embolism
  3. Cerebral venous thrombosis
  4. Venous thromboembolism in other sites
  5. Microvascular thrombosis
  6. Superficial venous thrombosis
  The following events defined and reported according to CTCAE v5.
  ii) Death
  iii) Composite clinical outcomes
  1. A composite of all thrombotic events: arterial, venous, microvascular and death.
  2. Major adverse cardiac and cerebrovascular events (MACCE)
  iv) Rate of change in cognitive function assessed by the Montreal Cognitive Assessment (MoCA) in conjunction with the Queen Square Cognitive Assessment score
B) Safety | 24 months
  (i) Bleeding: All bleeding events: major, clinically relevant non-major or minor (ii) Serious adverse events other than major bleeding (iii) Cerebral microbleeds (CMB) assessed with susceptibility-weighted imaging (SWI) as a surrogate marker of bleeding risk.
C) Health Economics | 24 months
  1. Quality of life (QoL) assessed using EQ-5D-5L
  2. Health and social care resource use assessed using trial follow-up visit case report forms (CRFs)
  3. Mean incremental cost per quality adjusted life year (QALY)
  Serious adverse events other than major bleeding using the criteria within the CTCAE version 5.
D) Anticoagulation intensity | 24 months
  1. Rivaroxaban i) Rivaroxaban anti-Xa levels
  2. Warfarin i) Time in target therapeutic range (TTR) ii) Amidolytic factor X as a lupus anticoagulant independent assessment of warfarin anticoagulant effect
ii) Changes in total brain volume, white matter volume and grey matter volume on T1w volumetric images on MRI | 24 Months
  This will be used as a marker for neurological efficacy of the IMP compared with current standard of care.

OTHER OUTCOMES:
E. Exploratory Outcomes | 24 months
  1. Rivaroxaban pharmacokinetic (PK) modelling
  2. Cerebral blood flow (CBF) derived from MR perfusion imaging using an arterial spin labelling (ASL) technique

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Cohen, Principal Investigator — University College London Hospitals NHS Foundation Trust/University College London
Locations (6):
- United Kingdom (6):
  - Epsom and St Helier University Hospitals NHS Trust, Epsom
  - Barts and the London Hospitals, Barts Health NHS Trust, London
  - Hammersmith Hospital, Imperial College Healthcare NHS Trust, London
  - Kings College Hospital NHS Foundation Trust, London
  - University College Hospitals NHS Foundation Trust, London
  - Queens Hospital, Barking, Havering and Redbridge University Hospitals NHS Trust, Romford

IPD SHARING:
Plan to Share IPD: No